CLINICAL TRIAL: NCT05020795
Title: Effect of Proximal Blood Flow Arrest During Endovascular Thrombectomy
Acronym: ProFATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21DI004
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Occlusion, Cerebrovascular
Keywords: Stroke; Large vessel occlusion; Balloon guide catheter; Flow arrest; Mechanical thrombectomy; Endovascular thrombectomy
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon inflation (Experimental): Endovascular thrombectomy with simultaneous balloon inflation using a balloon guide catheter
  Interventions: Procedure: Endovascular thrombectomy
- No balloon inflation (Active Comparator): Endovascular thrombectomy without simultaneous balloon inflation using a balloon guide catheter
  Interventions: Procedure: Endovascular thrombectomy

INTERVENTIONS:
Procedure: Endovascular thrombectomy — Clot retrieval for large vessel occlusion in acute ischaemic stroke

SUMMARY:
Endovascular thrombectomy (EVT) has become the standard of care for large vessel occlusion in acute ischaemic stroke (AIS). During clot-retrieval, simultaneous balloon inflation within the internal carotid artery offers transient proximal blood flow arrest, potentially preventing distal clot migration or embolisation to new vascular territories. Retrospective studies indicate that this may improve complete vessel recanalisation rates and may translate to improved functional independence. However, lack of high-quality evidence demonstrating the efficacy of simultaneous balloon inflation has led to clinical equipoise with heterogeneity of practice globally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute ischemic stroke presenting with a neurological deficit of (NIHSS ≥2)
* Intracranial arterial occlusion of the distal internal carotid artery or middle cerebral artery (M1/M2 segments) demonstrated with on clinical neuroimaging such as: computed tomography angiogram (CTA), magnetic resonance imaging angiogram (MRA), or digital subtraction angiography (DSA).
* ASPECTS score of >4 or by locally accepted ischaemic core/penumbra mismatch using computed tomography perfusion or magnetic resonance (CTP or MR) imaging.
* modified Rankin Scale, mRS<3
* Intention to treat with aspiration only or combination technique of stent-retriever + aspiration in the first pass attempt during endovascular thrombectomy

Exclusion Criteria:

* Severe stenosis (>90%), or tandem occlusion of the ipsilateral extracranial internal carotid artery.
* Previously deployed stents in the ipsilateral internal carotid artery.
* Dissections of the ipsilateral internal carotid artery.
* Unlikely to be available for 90 days follow-up (e.g. no fixed home address, visitor from overseas).
* Subject participating in a study involving an investigational drug or device that would impact this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Modified thrombolysis in cerebral infarction (mTICI) score of 2c-3 | Immediately after endovascular thrombectomy
  Near complete-complete vessel recanalisation

SECONDARY OUTCOMES:
Modified thrombolysis in cerebral infarction (mTICI) score of 2b-3 | Immediately after endovascular thrombectomy
  Successful vessel recanalisation
First pass effect (mTICI2c-3) | During endovascular thrombectomy procedure
  Near complete-complete vessel recanalisation after the first pass attempt at clot retrieval
New or distal vascular territory clot embolisation | Immediately after endovascular thrombectomy
Modified Rankin Scale 0-2 | 90 days
  Good functional outcome based on the modified Rankin scale of disability
Symptomatic intracranial haemorrhage | 24 hours after Endovascular thrombectomy
National Institutes of Health of Stroke Scale (NIHSS) | 24 hours
  Change in stroke severity
Mortality | 90 days
Total number of passes at clot retrieval | Immediately after endovascular thrombectomy
Procedure related complications | Immediately after endovascular thrombectomy
Total procedural time | Immediately after endovascular thrombectomy

CONTACTS AND LOCATIONS:
Overall Officials: Permesh Singh Dhillon, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Dhillon PS, Butt W, Podlasek A, Bhogal P, Lynch J, Booth TC, McConachie N, Lenthall R, Nair S, Malik L, Goddard T, Carraro do Nascimento V, Barrett E, Jethwa K, Krishnan K, Dineen RA, England TJ; ProFATE Investigators. Effect of Proximal Blood Flow Arrest During Endovascular Thrombectomy (ProFATE): A Multicenter, Blinded-End Point, Randomized Clinical Trial. Stroke. 2025 Feb;56(2):371-379. doi: 10.1161/STROKEAHA.124.049715. Epub 2024 Dec 19. PMID 39697177
- [Derived] Dhillon PS, Butt W, Podlasek A, Bhogal P, McConachie N, Lenthall R, Nair S, Malik L, Lynch J, Goddard T, Barrett E, Krishnan K, Dineen RA, England TJ. Effect of proximal blood flow arrest during endovascular thrombectomy (ProFATE): Study protocol for a multicentre randomised controlled trial. Eur Stroke J. 2023 Jun;8(2):581-590. doi: 10.1177/23969873231166194. Epub 2023 Mar 30. PMID 37231682